CLINICAL TRIAL: NCT01445327
Title: A Pilot Study of Markers of Tumor Burden and Radiation Toxicity in the Blood, Urine, and Stool of Patients Receiving Radiotherapy for Gastrointestinal Malignancies
Brief Title: Predictors of Tumor Response and of Radiation Therapy Side Effects in Patients With Gastrointestinal Cancers
Status: Terminated | Type: Observational
Why Stopped: Slow, insufficient accrual.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Deborah Citrin, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 070111; 07-C-0111; NCT00452946 (obsolete NCT alias)
Record Dates: First submitted 2011-09-30; First posted 2011-10-03 (Estimated); Results first posted 2022-02-01 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Esophageal Cancer; Stomach Cancer; Pancreatic Cancer
Keywords: Blood; Urine; Stool; Tumor Marker; Radiation Therapy; Gastrointestinal Cancer; Esophageal Cancer; Stomach; Pancreatic Cancer
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms; Pancreatic Neoplasms; Gastrointestinal Neoplasms | interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 10 cc in one ethylenediamine tetraacetic acid (EDTA) tube for plasma for Transforming growth factor beta 1 (TGFbeta1); 24cc total in serum separator tube (SST) for serum for extra-cellular markers; Stool - at least 10 gram (gm) in a sterile collection cup (leukocyte markers); Urine - at least 15 cubic centimeter (cc) in a sterile collection cup
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Markers of Tumor Burden and Radiation Toxicity: Serum, plasma, urine, and stool samples will be collected prior to radiotherapy for participants with gastrointestinal malignancies.
  Interventions: Other: Specimen collection

INTERVENTIONS:
Other: Specimen collection

SUMMARY:
Background:

* Gastrointestinal cancers are among the most commonly diagnosed cancers in the United States.
* There are currently no tests to predict how patients with gastrointestinal cancers will respond to radiation therapy or which patients may develop side effects from treatment.
* Studies on tumor cells in the stool, urine, or blood from patients may provide valuable information that can be used to develop tests to determine which patients may need more or less aggressive therapy.
* Studies of other substances in the stool, urine, or blood from patients may provide valuable information that can be used to develop tests to determine which patients are likely to develop side effects from radiation treatments.

Objectives:

* To collect blood, urine and stool specimens from patients with gastrointestinal cancers who will undergo radiation therapy.
* To study hormone and protein changes in these blood, urine and stool specimens before, during and after radiation treatment in order to develop a way to predict how gastrointestinal cancers will respond to radiation therapy and if patients with these cancers will develop side effects from radiation treatment.

Eligibility:

-Patients 18 years of age and older with cancer of the gastrointestinal tract (esophagus, stomach, pancreas, rectum) who plan to receive radiotherapy to the site of the cancer on an National Cancer Institute (NCI) protocol

Design:

Participants undergo the following procedures:

* Tumor biopsy: Before any treatment or at the time of surgery if it is the first treatment
* Urine collection: Before, during, and after treatment and at follow-up visits.
* Stool collection: Before, during, and after treatment and at follow-up visits.
* Blood collection: Before, during, and after treatment and at follow-up visits.
* Intestinal permeability assessment: Before any treatment, before radiation (if radiation is not the first treatment), 1 month after radiation is completed, and 3 months after radiation is completed. This test determines how the patients intestines are working to absorb sugar and may provide information about side effects from radiation treatments. Patients fast after midnight, then drink a small glass of sugars, and then do a 6-hour urine collection.

DETAILED DESCRIPTION:
Background:

* Gastrointestinal (GI) carcinomas represent one of the most commonly diagnosed malignancies in the United States.
* A sensitive and specific marker of tumor persistence or recurrence would permit a more accurate determination of the appropriateness of adjuvant therapy in patients with no clinical evidence of disease following curative resection and allow the diagnosis of recurrences at earlier stages that may be amenable to curative salvage therapies.
* A biomarker detectable shortly after treatment or in the early stages of chronic radiation toxicity may allow the identification of patients at risk and early intervention.

Objectives:

* Our primary objective is to determine if patient specific tumor markers in stool, urine, or serum can be reliably detected prior to treatment and followed after treatment to monitor the extent of residual disease.
* A second objective is to evaluate the predictive value of potential markers of chronic gastrointestinal injury after radiotherapy.

Eligibility:

* Age greater than or equal to 18 years
* Histologically confirmed carcinoma of the gastrointestinal tract (esophagus, stomach, pancreas, rectum)
* Planned to receive radiotherapy to the site of the gastrointestinal malignancy on an National Cancer Institute (NCI) protocol

Design:

* This protocol provides a means of acquiring tissue, serum, urine, and stool samples from patients who will receive radiation therapy as part of their treatment for gastrointestinal malignancies.
* Patients treated with radiation therapy on NCI treatment protocols will be asked to provide samples prior to any local or systemic therapy as well as before, during and after their radiation treatment.
* These samples will be tested for the presence of tumor specific deoxyribonucleic acid (DNA) mutations and aberrant methylation patterns determined to be present in each patient's tumor by screening of initial biopsy or surgical material.
* Tumor markers specific to each patient, such as tumor specific DNA mutations or aberrant DNA methylation, may provide an individualized method to evaluate disease status and determine prognosis after therapy. Additionally, a number of stool and serum markers will be explored as early indicators of acute and eventual chronic gastrointestinal injury in patients receiving radiotherapy to the abdomen.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age greater than or equal to 18 years.
* Histologically confirmed carcinoma of the gastrointestinal tract (esophagus, stomach, pancreas, bile duct, rectum).
* Treatment plan includes radiotherapy to the site of the gastrointestinal malignancy on an National Cancer Institute (NCI) protocol.
* Paraffin embedded tumor tissue from biopsy or surgery adequate in amount to perform polymerase chain reaction (PCR) and methylation specific PCR or willingness to undergo re-biopsy.

EXCLUSION CRITERIA:

* Inability to provide informed consent.
* Patients who have a history of prior therapeutic radiation.
* Patients with evidence of distant metastases on initial staging evaluation.
* Patients with other cancers excluding non-melanomatous skin cancers or carcinoma in situ.
* History of inflammatory bowel disease.
* History of collagen vascular disease or disease of altered collagen metabolism (end stage renal disease or hepatic fibrosis due to chronic hepatitis).
* History of hypersensitivity to radiation or a history of a disease which results in mucosal or other hypersensitivity to radiation (Ataxia-Telangiectasia, Bloom's Syndrome, Human Immunodeficiency Virus, Fanconi anemia, nevoid basal cell carcinoma syndrome, Li-Fraumeni syndrome, and Nijmegen breakage syndrome).
* Inability to return for follow-up visits.
* Patients who have previously received or are currently receiving MDX-101 (ipilimumab).
* Diagnosis of human immunodeficiency virus (HIV), Hepatitis B, or Hepatitis C.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with gastrointestinal tumors that will receive radiation therapy at the National Institutes of Health (NIH) Clinical Center as part of their treatment.
Sampling Method: Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2007-02-20 (Actual); Primary Completion 2014-05-22 (Actual); Study Completion 2014-05-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah E Citrin, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jemal A, Siegel R, Ward E, Murray T, Xu J, Smigal C, Thun MJ. Cancer statistics, 2006. CA Cancer J Clin. 2006 Mar-Apr;56(2):106-30. doi: 10.3322/canjclin.56.2.106. PMID 16514137
- [Background] Seamonds B, Yang N, Anderson K, Whitaker B, Shaw LM, Bollinger JR. Evaluation of prostate-specific antigen and prostatic acid phosphatase as prostate cancer markers. Urology. 1986 Dec;28(6):472-9. doi: 10.1016/0090-4295(86)90146-9. PMID 2431533
- [Background] Guillet J, Role C, Duc AT, Francois H. Prostate-specific antigen (PSA) in the management of 500 prostatic patients. Am J Clin Oncol. 1988;11 Suppl 2:S61-2. doi: 10.1097/00000421-198801102-00013. PMID 2468274

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants With Esophageal Cancer Treated With 4680-5040 Centigray (cGy) Total Dose + Chemotherapy: Serum, plasma, urine, and stool samples will be collected prior to radiotherapy for participants with gastrointestinal malignancies.
  Participants with esophageal cancer received 4680-5040 cGy total dose, generally with concurrent chemotherapy (cisplatin and Fluorouracil (5-FU). Treatment cycles varied by participant.
- Participants With Pancreatic Cancer Treated With 5400 Centigray (cGy) + Xeloda: Serum, plasma, urine, and stool samples will be collected prior to radiotherapy for participants with gastrointestinal malignancies.
  Participants with pancreatic cancer received 5400 cGy with Xeloda. Treatment cycles varied by participant.
- Participants With Rectal Cancer Treated With 5040 Centigray (cGy) With Concurrent Xeloda: Serum, plasma, urine, and stool samples will be collected prior to radiotherapy for participants with gastrointestinal malignancies.
  Participants with rectal cancer received 5040 cGy with concurrent Xeloda. Treatment cycles varied by participant.
Period: Overall Study
Arm/Group | Participants With Esophageal Cancer Treated With 4680-5040 Centigray (cGy) Total Dose + Chemotherapy | Participants With Pancreatic Cancer Treated With 5400 Centigray (cGy) + Xeloda | Participants With Rectal Cancer Treated With 5040 Centigray (cGy) With Concurrent Xeloda
Started | 3 | 1 | 5
Completed | 3 | 1 | 5
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Participants With Esophageal Cancer Treated With 4680-5040 Centigray (cGy) Total Dose + Chemotherapy | Participants With Pancreatic Cancer Treated With 5400 Centigray (cGy) + Xeloda | Participants With Rectal Cancer Treated With 5040 Centigray (cGy) With Concurrent Xeloda | Total
Number analyzed (Participants) | 3 | 1 | 5 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 0 | 5 | 7
  >=65 years | 1 | 1 | 0 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.55 (14.19) | 69 (0) | 54.75 (2.96) | 61.76 (8.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 3 | 4
  Male | 2 | 1 | 2 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 1 | 5 | 9
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1
  White | 3 | 1 | 4 | 8
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 1 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Specific Tumor Markers in Stool, Urine, or Serum Detected Prior to Treatment and After Treatment
Description: Here are the number of participants with specific tumor markers in stool, urine, or serum detected prior to treatment and after treatment to monitor the extent of residual disease.
Time Frame: Prior to treatment (baseline) and after treatment, up to 19 months
Population: A minimum of 120 participants must be enrolled to perform analyses to determine specific tumor markers in stool, urine for this outcome measure. Because the study was prematurely terminated due to slow, insufficient accrual and requirements for enrolment, assays were not performed on the collected samples, thus no data is reported for this outcome measure. It would be inappropriate to report an analysis for this outcome measure based on the enrollment of 9 participants.
Arm/Group | Participants With Esophageal Cancer Treated With 4680-5040 Centigray (cGy) Total Dose + Chemotherapy | Participants With Pancreatic Cancer Treated With 5400 Centigray (cGy) + Xeloda | Participants With Rectal Cancer Treated With 5040 Centigray (cGy) With Concurrent Xeloda
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Number of Participants With Chronic Gastrointestinal Injury After Radiotherapy
Description: Gastrointestinal injury after radiotherapy is influenced by radiation dose (i.e. radiation toxicity) delivered to abdominal organs and can result in gastrointestinal radiation toxicity. Early detection of radiation toxicity (i.e. inflammation, fibrosis) may lead to a good outcome for a participant and late detection and radiation toxicity in the intestinal wall may lead to a bad outcome for a participant.
Time Frame: After radiotherapy, up to 19 months
Population: A minimum of 120 participants must be enrolled to perform analyses to determine gastrointestinal injury for this outcome measure. Because the study was prematurely terminated due to slow, insufficient accrual, and requirements for enrolment, analyses were not performed, and no data is reported for this outcome measure. It would be inappropriate to report an analysis for this outcome measure based on the enrollment of 9 participants.
Arm/Group | Participants With Esophageal Cancer Treated With 4680-5040 Centigray (cGy) Total Dose + Chemotherapy | Participants With Pancreatic Cancer Treated With 5400 Centigray (cGy) + Xeloda | Participants With Rectal Cancer Treated With 5040 Centigray (cGy) With Concurrent Xeloda
Number analyzed (Participants) | 0 | 0 | 0

3. Other Pre Specified Outcome: Here is the Number of Participants With Serious and Non-serious Adverse Events Assessed by the Common Toxicity Criteria (CTC) v3.0.
Description: Here is the number of participants with serious and non-serious adverse events assessed by the Common Toxicity Criteria (CTC) v3.0. A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, an average of 19 months
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Esophageal Cancer Treated With 4680-5040 Centigray (cGy) Total Dose + Chemotherapy | Participants With Pancreatic Cancer Treated With 5400 Centigray (cGy) + Xeloda | Participants With Rectal Cancer Treated With 5040 Centigray (cGy) With Concurrent Xeloda
Number analyzed (Participants) | 3 | 1 | 5
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, an average of 19 months.
Arm/Group | Participants With Esophageal Cancer Treated With 4680-5040 Centigray (cGy) Total Dose + Chemotherapy | Participants With Pancreatic Cancer Treated With 5400 Centigray (cGy) + Xeloda | Participants With Rectal Cancer Treated With 5040 Centigray (cGy) With Concurrent Xeloda
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/1 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/1 | 0/5
Other Adverse Events (participants affected / at risk) | 0/3 | 0/1 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2007-02-11): https://cdn.clinicaltrials.gov/large-docs/27/NCT01445327/Prot_SAP_ICF_000.pdf